CLINICAL TRIAL: NCT01424228
Title: A Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Quality of Life, Safety and Tolerability of Long-term Treatment (24 Weeks) With Prucalopride in Subjects Aged ≥18 Years With Chronic Constipation
Brief Title: Evaluation of Long-term Prucalopride Treatment With Chronic Constipation in Subjects Aged ≥ 18 Years
Acronym: SPD555-401
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M0001-C401; 2011-000670-62 (EudraCT Number); SPD555-401 (Other: Shire)
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Constipation
Keywords: Long term; Constipation; Digestive signs and symptoms
MeSH Terms: conditions — Constipation; Signs and Symptoms, Digestive | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 2 mg tablet once daily before breakfast
  Interventions: Drug: placebo
- prucalopride (Active Comparator): Prucalopride 2 mg once daily before breakfast
  Interventions: Drug: prucalopride

INTERVENTIONS:
Drug: placebo — Placebo matching tablet 2 mg once daily before breakfast for 24 weeks
  Arms: Placebo
Drug: prucalopride — Prucalopride 2 mg daily before breakfast
  1 mg for subjects >65 years; in case of insufficient response 2 mg at week 2 or week 4
  Arms: prucalopride

SUMMARY:
The purpose of this trial is to evaluate the long-term (24 weeks) efficacy of prucalopride versus placebo in subjects aged 18 years and older with chronic constipation.

DETAILED DESCRIPTION:
In this phase IV trial a total of 340 subjects (170 subjects per treatment group), with chronic constipation, are planned to be randomly assigned to double-blind treatment.

The trial duration for a subject can be 26 to 28 weeks in total, including a 2- to 4-week run-in phase followed by a 24-week double-blind treatment phase. The patient will complete an e-diary.

Adult subjects (≥18 to <65 years of age) will take 2 mg prucalopride or matching placebo throughout the entire 24-week treatment period. Elderly subjects (≥65 years of age) will start at a dose of 1 mg prucalopride or matching placebo. In case of insufficient response the daily dose has to be increased to 2 mg (i.e. changed to 2 mg prucalopride or matching placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant, non-breastfeeding female out-patient ≥18 years of age (no upper age limit).
2. Subject has a history of constipation. The subject reports an average of ≤2 SBM/week that result in a feeling of complete evacuation (SCBM).
3. Subject agrees to stop his/her current laxative treatment and is willing to use rescue medication according to the rescue rule [bisacodyl/enemas].

Exclusion Criteria:

1. Subjects in whom constipation is thought to be drug-induced
2. Subjects using any disallowed medication.
3. Subjects who previously used prucalopride.
4. Subjects suffering from secondary causes of chronic constipation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2011-04-06 (Actual); Primary Completion 2012-12-19 (Actual); Study Completion 2012-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (60):
- Belgium (4):
  - Universitaire Ziekenhuizen Leuven, Leuven, Flemish Brabant
  - Cliniques Universitaires St. Luc, Brussels
  - Huisartspraktijk Jaak Mortelmans, Ham
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège
- Czechia (7):
  - Fakultní Thomayerova nemocnice s poliklinikou, Praha 4 - Krc, Prague
  - Derma Plus s.r.o., České Budějovice
  - Oblastní nemocnice Kolín, a.s., Kolín
  - Diagnostika a Lécba Zažívacích Chorob, s.r.o., Ostrava-Hrabuvka
  - MONSE s.r.o, Prague
  - Nemocnice Tábor, a.s., Tábor
  - Orlickoústecká Nemocnice a.s, Ústí nad Orlicí
- Hungary (14):
  - Békés Megyei Képviselotestület Pándy Kálmán Kórháza, Gyula, Bekes County
  - Szegedi Tudományegyetem I. Sz. Belgyógyászati Klinika, Szeged, Csongrád megye
  - Dr. Bugyi István Kórház, Szentes, Csongrád megye
  - Petz Aladár Megyei Oktató Kórház, Győr, Győr-Moson-Sopron
  - Karolina Kórház Rendelointézet, Mosonmagyaróvar, Győr-Moson-Sopron
  - Fejér Megyei Szent György Kórház, Székesfehérvár, Pejer
  - Fundamed Háziorvosi Szövetkezet, Érd, Pest County
  - UNO Medical Trials, Kft., Budapest
  - Pannónia Magánorvosi Centrum Kft., Budapest
  - BAZ Megyei és Egyetemi Oktató Kórház, Miskolc
  - Clinfan Kft. SMO, Szekszárd
  - CRU Hungary Kft., Szikszó
  - Bíró Praxis Kft., Úrhida
  - Jávorszky Ödön Városi Kórház, Vác
- Italy (6):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedale San Martino, Genova
  - Policlinico Universitario, Padua
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Policlinico Universitario Campus Biomedico, Roma
  - Azienda Policlinico Umberto I di Roma, Roma
- Poland (6):
  - Krakowskie Centrum Medyczne NZOZ, Krakow, Lesser Poland Voivodeship
  - Przychodnia Polskiej Fundacji Gastroenterologii Filia Nr 1 NZOZ, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki w Opolu, Opole, Opole Voivodeship
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Centrum Medyczne sw. Lukasza Sp. z o.o., Częstochowa, Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej "SONOMED", Szczecin, West Pomeranian Voivodeship
- Romania (11):
  - Spitalul Militar Central Bucuresti, Bucharest, București
  - Centrul Medical Sana, Bucharest, București
  - Spitalul Clinic Judetean Cluj,Clinica Medicala I, Cluj-Napoca, Cluj
  - Biomed Plus SRL, Craiova, Dolj
  - SC Cabinet Medical Dr. Blaj Stefan SRL, Bucharest, Sector 5
  - Centrul Medical Tuculanu SRL, Timișoara, Timiș County
  - Endocenter Medicina Integrativa SRL, Bucharest
  - Gastromedica SRL, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - CMI de Gastroenterologie Dobru Daniela, Târgu Mureş
  - Policlinic Algomed SRL, Timișoara
- Slovakia (6):
  - Lama Medical Care s.r.o., Gastroentero-hepatologicke centrum Thalion, Bratislava
  - Gastroenterologická ambulancia, Košice
  - PIGEAS s.r.o., Martin
  - Radvanská lekáren, spol. s r.o.,, Nitra
  - Gastro I.s.r.o., Prešov
  - GEA s.r.o Gastroenterologicka ambulancia, Trnava
- Spain (3):
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Nuestra Señora de Valme, Seville
- Sweden (3):
  - Sahlgrenska Universitetsjukhuset, Gothenburg, Västra Götaland County
  - Aleris Specialistvård Sabbatsberg, Stockholm
  - Karolinska University Hospital Solna, Stockholm

REFERENCES:
- [Derived] Lembo A, Staller K, Boules M, Feuerstadt P, Spalding W, Gabriel A, Youssef A, Xie Y, Terreri B, Cash BD. Efficacy and safety of prucalopride in patients with chronic idiopathic constipation stratified by age, body mass index, and renal function: a post hoc analysis of phase III and IV, randomized, placebo-controlled clinical studies. Therap Adv Gastroenterol. 2024 Dec 10;17:17562848241299731. doi: 10.1177/17562848241299731. eCollection 2024. PMID 39664231
- [Derived] Staller K, Hinson J, Kerstens R, Spalding W, Lembo A. Efficacy of Prucalopride for Chronic Idiopathic Constipation: An Analysis of Participants With Moderate to Very Severe Abdominal Bloating. Am J Gastroenterol. 2022 Jan 1;117(1):184-188. doi: 10.14309/ajg.0000000000001521. PMID 34585675
- [Derived] Piessevaux H, Corazziari E, Rey E, Simren M, Wiechowska-Kozlowska A, Kerstens R, Cools M, Barrett K, Levine A. A randomized, double-blind, placebo-controlled trial to evaluate the efficacy, safety, and tolerability of long-term treatment with prucalopride. Neurogastroenterol Motil. 2015 Jun;27(6):805-15. doi: 10.1111/nmo.12553. Epub 2015 Mar 25. PMID 25808103

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Tablet once daily before breakfast
- Prucalopride: 1 mg or 2 mg tablet once daily before breakfast
Period: Overall Study
Arm/Group | Placebo | Prucalopride
Started | 182 | 182
Completed | 126 | 135
Not Completed | 56 | 47
Not completed — Withdrawal by Subject | 27 | 11
Not completed — Adverse Event | 10 | 14
Not completed — Sponsor's decision | 9 | 12
Not completed — Lack of Efficacy | 5 | 7
Not completed — inclusion/exclusion criteria not met | 2 | 2
Not completed — Non-compliance | 2 | 0
Not completed — Worsening of symptoms | 1 | 0
Not completed — Unplanned journey | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was used for demographics. The Safety Population includes all subjects randomized into the study who took at least 1 dose of investigational product. Three subjects did not receive investigational product and therefore were not included in the Safety Population (n = 361).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Prucalopride | Total
Number analyzed (Participants) | 180 | 181 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (16.25) | 49.4 (15.78) | 48.9 (16.00)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 149 | 146 | 295
  > = 65 years to <75 years | 20 | 26 | 46
  >=75 years | 11 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 155 | 308
  Male | 27 | 26 | 53
Region of Enrollment [Count of Participants; unit: Participants] — This includes all randomized subjects (n = 364).
  Participants
    Romania | 38 | 37 | 75
    Poland | 34 | 31 | 65
    Hungary | 29 | 31 | 60
    Slovakia | 28 | 29 | 57
    Italy | 19 | 18 | 37
    Spain | 11 | 8 | 19
    Belgium | 8 | 11 | 19
    Sweden | 9 | 9 | 18
    Czech Republic | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With an Average of ≥3 Spontaneous Complete Bowel Movements (SCBM) Per Week Over the 24 Week Treatment Period
Description: Spontaneous Bowel Movements defined as a bowel movement that is not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.
Time Frame: Over 24 week treatment period
Population: Intent-to-Treat Population (ITT) includes all subjects randomized into the study who took at least 1 dose of investigational product. There were 21 subjects with a risk of potential unblinding due to an error in the randomization system who were excluded from the ITT Population to avoid the risk of bias to the study results.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 169 | 171
percentage of subjects | 20.7 | 25.1
Statistical Analysis 1: Comparison: Placebo vs Prucalopride; Test type: Superiority or Other; p = 0.367, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Subjects With an Increase of ≥1 Spontaneous Complete Bowel Movement (SCBM) Per Week Up to 24 Weeks
Time Frame: Over 24 week treatment period
Population: Intent-to-Treat Population (ITT) includes all subjects randomized into the study who took at least 1 dose of investigational product. The 21 subjects with a risk of potential unblinding due to an error in the randomization system were excluded from the ITT Population to avoid the risk of bias to the study results.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 169 | 171
percentage of subjects | 42.0 | 48.0

3. Secondary Outcome: Average Number of Spontaneous Complete Bowel Movements (SCBM) Per Week Up to 24 Weeks
Time Frame: Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: SCBM/week
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 165 | 158
SCBM/week | 1.7 (1.86) | 2.1 (1.96)

4. Secondary Outcome: Change From Baseline in Spontaneous Complete Bowel Movements Per Week at Up to 24 Weeks
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: SCBM/week
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 165 | 158
SCBM/week | 1.3 (1.77) | 1.7 (1.90)

5. Secondary Outcome: Percent of Subjects With an Average Weekly Frequency of at Least 3 SCBM by Week
Time Frame: Over 24 week treatment period
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 169 | 171
percentage of subjects
  Week 1 | 18.3 | 32.2
  Week 2 | 23.1 | 34.5
  Week 3 | 22.5 | 32.2
  Week 4 | 23.1 | 31.6
  Week 5 | 26.6 | 27.5
  Week 6 | 28.4 | 29.2
  Week 7 | 29.0 | 29.8
  Week 8 | 26.0 | 30.4
  Week 9 | 27.8 | 33.3
  Week 10 | 26.0 | 30.4
  Week 11 | 25.4 | 37.4
  Week 12 | 27.2 | 33.9
  Week 13 | 23.7 | 30.4
  Week 14 | 30.2 | 35.7
  Week 15 | 24.9 | 29.2
  Week 16 | 29.6 | 35.1
  Week 17 | 28.4 | 35.1
  Week 18 | 30.2 | 32.7
  Week 19 | 32.0 | 32.2
  Week 20 | 24.9 | 37.4
  Week 21 | 26.6 | 30.4
  Week 22 | 27.8 | 32.7
  Week 23 | 30.2 | 31.0
  Week 24 | 32.0 | 31.6

6. Secondary Outcome: Percent of Subjects With an Average Weekly Frequency of at Least 3 SCBM by 4-Week Treatment Period
Time Frame: Over 24 week treatment period
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 169 | 171
percentage of subjects
  First 4-week period | 18.3 | 26.9
  Second 4-week period | 23.7 | 25.7
  Third 4-week period | 23.7 | 29.2
  Fourth 4-week period | 22.5 | 29.2
  Fifth 4-week period | 23.7 | 33.3
  Sixth 4-week period | 24.9 | 26.9

7. Secondary Outcome: Change From Baseline in Average Consistency Per SCBM at Up to 24 Weeks
Description: Consistency measured using the 7-point Bristol scale where 1-2 indicate constipation (=hard/very hard), 3-4 are ideal stools (=normal), and 5-7 tending toward diarrhea.
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 67 | 55
units on a scale | -0.1 (1.79) | -0.1 (1.31)

8. Secondary Outcome: Change From Baseline in Percent SCBM With a Consistency of Normal and Hard/Very Hard at Up to 24 Weeks
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of SCBM
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 67 | 55
percentage of SCBM
  Normal consistency | 16.82 (42.365) | 25.71 (40.1)
  Hard/Very Hard consistency | -9.11 (41.495) | -13.82 (31.349)

9. Secondary Outcome: Change From Baseline in Straining Per SCBM at Up to 24 Weeks
Description: Straining was evaluated on a 5-point scale (0=none, 1=mild, 2=moderate, 3=severe, or 4=very severe)
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 67 | 55
units on a scale | -0.44 (0.948) | -0.23 (0.870)

10. Secondary Outcome: Change From Baseline in Percent SCBM With No Straining and Severe/Very Severe Straining at Up to 24 Weeks
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of SCBM
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 67 | 55
percentage of SCBM
  No straining | 11.14 (39.786) | 6.61 (33.916)
  Severe/Very Severe straining | -9.85 (29.711) | -4.49 (28.177)

11. Secondary Outcome: Change From Baseline in Percent SBM With Sensation of Complete Evacuation at Up to 24 Weeks
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of SBM
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 149 | 138
percentage of SBM | 20.94 (32.619) | 24.22 (32.878)

12. Secondary Outcome: Time to First SCBM After Investigational Product Intake on Day 1 and Day 28
Time Frame: Day 1 and 28
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 169 | 171
hours
  Day 1 | 359.67 [179.6 to 461.42] | 100.83 [74.0 to 170.75]
  Day 28 | 100.58 [75.2 to 199.02] | 81.78 [52.25 to 151.05]

13. Secondary Outcome: Change From Baseline in the Number of Bisacodyl Tablets Taken Per Week at Up to 24 Weeks
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: tablets/week
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 140 | 144
tablets/week | -0.68 (1.583) | -0.97 (1.821)

14. Secondary Outcome: Change From Baseline in the Number of Days With Rescue Medication Taken Per Week at Up to 24 Weeks
Description: Rescue medications include laxatives and enemas.
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 140 | 144
days/week | -0.42 (0.892) | -0.54 (1.018)

15. Secondary Outcome: Change From Baseline in the Patient Assessment of Constipation - Symptom (PAC-SYM) Questionnaire Score at Up to the Final On Treatment Assessment Value
Description: The PAC-SYM is a validated 12-item questionnaire for the evaluation of severity of symptoms of constipation in subjects with constipation. Items are rated on a 5-point Likert scale: 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. Total score ranges from 0 to 48. Lower scores indicate improvement in symptoms. A 1-point improvement in PAC-SYM total score was considered clinically meaningful.
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 167 | 167
units on a scale | -0.68 (0.929) | -0.55 (0.794)

16. Secondary Outcome: Change From Baseline in the Patient Assessment of Constipation - Quality of Life (PAC-QOL) Score at Up to the Final On Treatment Assessment Value
Description: The PAC-QOL is a validated 28-item questionnaire for the evaluation of quality of life in subjects with constipation. Items are rated on a 5-point Likert scale: 0=not at all/none of the time, 1=a little bit/a little bit of the time, 2=moderately/some of the time, 3=quite a bit/most of the time, 4=extremely/all of the time. Total score ranges from 0-112. Lower scores indicate improvement in symptoms. A 1-point improvement in PAC-QOL total score was considered clinically meaningful.
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 162 | 166
units on a scale | -0.73 (0.902) | -0.67 (0.932)

17. Secondary Outcome: Change From Baseline in the Short Form-36 Health Survey (SF-36) Score at Up to the Final On Treatment Assessment Value
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Total score ranges from 0 (lowest level of health) - 100 (highest level of health) on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability (i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability). Higher scores are associated with better quality of life.
Time Frame: Baseline and Over 24 week treatment period
Population: ITT population. Not all subjects in the ITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 164 | 167
units on a scale
  Mental component | 3.786 (10.0887) | 3.179 (10.5714)
  Physical component | 3.331 (6.9830) | 2.965 (6.9320)

ADVERSE EVENTS:
Description: The Safety Population includes all subjects randomized into the study who took at least 1 dose of investigational product. Three subjects did not receive investigational product and therefore were not included in the Safety Population (n = 361).
Arm/Group | Placebo | Prucalopride
Serious Adverse Events (participants affected / at risk) | 4/180 | 4/181
Other Adverse Events (participants affected / at risk) | 23/180 | 41/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=180) | Prucalopride (N=181)
Colitis ischemic (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischemic stroke (Nervous system disorders) | 1 | 0
Abnormal behavior (Psychiatric disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=180) | Prucalopride (N=181)
Abdominal pain (Gastrointestinal disorders) | 8 | 18
Nausea (Gastrointestinal disorders) | 7 | 13
Headache (Nervous system disorders) | 10 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.